CLINICAL TRIAL: NCT06460740
Title: Combined Effects of 4-7-8 Breathing Technique and Stationary Cycle on Physical Performance, Quality of Life and Dyspnea in Post CABG Patients
Brief Title: Comb Effect of 4-7-8 Breathing Technique and Stationary Cycle on PP, QOL and Dyspnea in Post CABG Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/47039 Samrah Mahmood
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Post-cardiac Surgery
Keywords: 4-7-8 breathing technique; stationary cycling; Post CABG; physical performance; quality of life; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only the patients will be blind its a single blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-7-8 breathing technique (Experimental): 4-7-8 breathing technique and stationary cycling
  Interventions: Other: 4-7-8 breathing technique
- Stationary cycling (Active Comparator): Stationary Cycling
  Interventions: Other: Stationary Cycling

INTERVENTIONS:
Other: 4-7-8 breathing technique — Treatment will be given 18 exercise sessions per month (four to five times per week). The patient at first will be directed to sit or lie down, in which manner they feel sense of comfort. Then they are asked to exhale completely through mouth emptying their lungs. Then closing their lips and inhaling silently through nose while counting on the count of 4 seconds, holding their breath for a count of 7 seconds and exhale slowly through semi-closed lips making a Whoosh sound for a count of 8 seconds. Inhale, hold breath, and exhale ratio of 4:7:8. In aerobic protocol, F (frequency) subjects will receive training up to 18 exercise sessions per month (four to five times per week). I (intensity) subjects will receive training up to intensity of 70 to 75 %, T & T (Time and Type) subjects will receive training up to 20 minutes of bicycling.
  Other Names: Generalized Active ROM
  Arms: 4-7-8 breathing technique
Other: Stationary Cycling — In aerobic protocol, F (frequency) subjects will receive training up to 18 exercise sessions per month (four to five times per week). I (intensity) subjects will receive training up to intensity of 70 to 75 %, T & T (Time and Type) subjects will receive training up to 20 minutes of bicycling
  Other Names: Generalized Active ROM
  Arms: Stationary cycling

SUMMARY:
To determine the combined effects of 4-7-8 breathing technique and stationary cycle on physical performance, quality of life and dyspnea in post CABG patients.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria and will be excluded from the exclusion criteria will be recruited by convenient sampling technique and will be allocated to simple randomization process. By taking a sample of 58 patients through non-probability convenience sampling and randomly assigning them into two groups, Group A and Group B for 18 exercise sessions per month (four to five times in a week), out of which group A will receive 4-7-8 breathing technique and stationary cycle (n=29). Group B will alone receive Stationary cycle (n=29). The study will be Single-blind where patients will be only blind. Pre and post treatment training outcomes of physical performance will be measured through 6-minute walk test, quality of life will be measured through Short-item 36 (SF-36) questionnaire 2.0 version and dyspnea will be measured through modified Borg scale. The data will be analyzed through SPSS version 26. Generalized active range of motion will be given to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a successful CABG (no complications during surgery
* and/or in the following weeks)
* Female and male whose age between 40 to 70 years of age
* Phase II cardiac rehab patients
* Patients who were extubated and hemodynamically stable
* Patients with stable chronic heart failure.
* Patients had no arrhythmias
* Patients who had ability to read and write
* Patients who voluntarily participated in the study.

Exclusion Criteria:

* Ventricular Septal defect repair.
* Patients have limitation of motion that prevents them from performing physical activities such as walking for 6 minute.
* Patients who had undergone previous cardiac surgery.
* Severe renal dysfunction requiring dialysis.
* Altered level of consciousness.
* A history of musculoskeletal problems
* Having an orthopedic problem that prevents the use of lower and upper extremity bikes.
* Cancer patients receiving radiotherapy and chemotherapy.
* Clinical diagnosis of uncontrolled Diabetes Mellitus and Hypertension.
* Physical Discomfort at any stage of the study and/or any reaction to the tests (nausea, dizziness, discomfort, feeling faint, tachycardia, excessive sweating), and if they failed to attend the scheduled sessions.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Physical Performance 6MWT | 4th week
  Changes from baseline The 6-minute walk test (6MWT) was developed by American Thoracic society and was officially introduced in 2002, coming along with a comprehensive guideline. The 6MWT is an easy, safe, reliable and simple cardiopulmonary sub maximal functional testing modality, used to assess functional capacity and to evaluate the cardiac and pulmonary rehabilitation treatment or intervention. (16) The individuals were requested to walk as far-off as they are able to on a smooth area for about 6 minutes. Individuals were permitted to take a rest or stop from walking if it was required then continue again as quick as they can. The distance covered by individuals for this test was measured in meters.

SECONDARY OUTCOMES:
SF-36 Quality of Life Questionnaire version 2.0 | 4th week
  Changes from baseline the 36 item Short-Form Survey (SF-36) is an outcome measure standardized structured questionnaire that is internationally and widely approved to evaluate the quality of life (QOL) of post CABG patients. The questionnaire was developed and used for collecting a data. The content validity was obtained from 7 experts. The questionnaire was found to be valid in assessing QOL. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Modified Borg Dyspnea Scale | 4th week
  Changes from baseline Borg rate of perceived exertion (RPE) or Rate of perceived dyspnea (RPD) is an outcome measuring scale was developed by Swedish researcher Gunnar Borg in the 1998, allowing the individuals to rate their level of exertion during exercise subjectively American College of Sports Medicine (ACSM), 2010. It is proposed for all patients who underwent and going through Rehabilitation and endurance training as well as used in research. It scores from 0 to 10, using numeric values to rate how much effort an activity takes or to rate the difficulty of breathing. The zero point in a scale, indicates breathing is causing no difficulty at all or no exertion at all progressing through to ten point where breathing difficult is at maximum point.

CONTACTS AND LOCATIONS:
Overall Officials: Qurat ul-Ain, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Medicare Cardiac and General Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wahdan Abd El-Aziz W, Attia Kandee N, Elsayed Mansour H. The Effect of Early SixMinute Walking Test Post-Coronary Artery Bypass Graft on Walking Tolerance and Physiological Parameters. Egyptian Journal of Health Care. 2020;11(3):784-94.
- [Background] Ambina K, Shalimol U, Anjana A. Quality of Life among Post CABG Patients. Prof(Dr) RK Sharma. 2020;20(4):41535.
- [Background] Abdelaziz Mohammed F, Shoeib Ali F. Effect of Early Ambulation Program on Selected Outcomes among Patients Undergoing Cardiac Surgery. Egyptian Journal of Health Care. 2022;13(4):888-904.
- [Background] Schulte B, Nieborak L, Leclercq F, Villafane JH, Sanchez Romero EA, Corbellini C. The Comparison of High-Intensity Interval Training Versus Moderate-Intensity Continuous Training after Coronary Artery Bypass Graft: A Systematic Review of Recent Studies. J Cardiovasc Dev Dis. 2022 Sep 28;9(10):328. doi: 10.3390/jcdd9100328. PMID 36286280
- [Background] Kansara P, Patel S. Effect of Post Operative Physiotherapy in Patients with CABG to Improve Cardiovascular Endurance-A Randomised Controlled Trial.
- [Background] Yükselmiş Ö. The Effect of Cycling and Arm Ergometer Exercises on Physical and Psychosocial Functions: Application in Patients Undergoing Coronary Artery Bypass Surgery. Open Journal of Therapy and Rehabilitation. 2022;10(2):39-53
- [Background] Munir U, Umar Riaz NF, Sahar W, Tariq K. Effects of Preoperative Aerobic Training for Improving Postoperative Functional Mobility in Coronary Artery Bypass Graft Patients. 2023.
- [Background] Naqvi M, Khan MS, Perwaiz S, Ibrahim Q, Khan MW, Khan TY. Comparative analysis on the efficacy of aerobic capacity in cardiac rehabilitation obese and non-obese phase ii patient. International Journal of Physiotherapy. 2019:64-9.
- [Background] Vierra J, Boonla O, Prasertsri P. Effects of sleep deprivation and 4-7-8 breathing control on heart rate variability, blood pressure, blood glucose, and endothelial function in healthy young adults. Physiol Rep. 2022 Jul;10(13):e15389. doi: 10.14814/phy2.15389. PMID 35822447
- [Background] Krasavina T, Zaborova V, Lazareva I, Yurku K, Putilo V, Gameeva V, et al. Rehabilitation of patients with coronary heart disease after coronary artery bypass grafting at the stationary stage. Journal of IMAB-Annual Proceeding Scientific Papers. 2023;29(2):4980-3.
- [Background] Hamed LA, Elsayed SM. Effect of Deep Breathing Exercises on Pain after Cardiac Catheterization: A Randomized Controlled Trial.
- [Background] Gambassi BB, Almeida FJF, Almeida AEAF, Ribeiro DAF, Gomes RSA, Chaves LFC, Sousa TMDS, Nina VJDS. Acute Response to Aerobic Exercise on Autonomic Cardiac Control of Patients in Phase III of a Cardiovascular Rehabilitation Program Following Coronary Artery Bypass Grafting. Braz J Cardiovasc Surg. 2019 Jun 1;34(3):305-310. doi: 10.21470/1678-9741-2019-0030. PMID 31310469
- [Background] Sheraz S, Ayub H, Ferraro FV, Razzaq A, Malik AN. Clinically Meaningful Change in 6 Minute Walking Test and the Incremental Shuttle Walking Test following Coronary Artery Bypass Graft Surgery. Int J Environ Res Public Health. 2022 Nov 1;19(21):14270. doi: 10.3390/ijerph192114270. PMID 36361150
- [Background] Moreira JMA, Grilo EN. Quality of life after coronary artery bypass graft surgery - results of cardiac rehabilitation programme. J Exerc Rehabil. 2019 Oct 28;15(5):715-722. doi: 10.12965/jer.1938444.222. eCollection 2019 Oct. PMID 31723562
- [Background] Ghorbani A, Hajizadeh F, Sheykhi MR, Mohammad Poor Asl A. The Effects of Deep-Breathing Exercises on Postoperative Sleep Duration and Quality in Patients Undergoing Coronary Artery Bypass Graft (CABG): a Randomized Clinical Trial. J Caring Sci. 2018 Dec 1;8(4):219-224. doi: 10.15171/jcs.2019.031. eCollection 2019 Dec. PMID 31915624
- [Background] Radi B, Ambari AM, Dwiputra B, Intan RE, Triangto K, Santoso A, Setianto B. Determinants and Prediction Equations of Six-Minute Walk Test Distance Immediately After Cardiac Surgery. Front Cardiovasc Med. 2021 Aug 19;8:685673. doi: 10.3389/fcvm.2021.685673. eCollection 2021. PMID 34490363